CLINICAL TRIAL: NCT05921019
Title: The Efficacy of Laser Acupuncture on the Diabetes-induced Peripheral Neuropathy: Basic and Clinical Research
Brief Title: Laser Acupuncture on Diabetes-induced Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taiwan Municipal An-Nan Hospital-China Medical University (Other)
Responsible Party: Principal Investigator, Yu Chen, Chiu, attending physician, Taiwan Municipal An-Nan Hospital-China Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANHRF111-06
Record Dates: First submitted 2023-06-15; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: diabetic peripheral neuropathy; laser acupuncture

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either the laser acupuncture, the sham laser acupuncture group using a block randomization method with allocation ratio of 1:1. According to the previous randomization assignment, each patient will be assigned to 2 groups: (1) the laser acupuncture group and (2) the sham laser acupuncture group. Only the statistician is aware of the randomized order for each participant. Each participant will receive 24 interventions within 8 weeks, including three interventions per week for 8 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: Before study commencement, the statistician created a randomization sequence using IBM® SPSS® Statistics and contained it in sealed envelopes. The balanced sample size was ensured by dividing the participants into blocks of two. All eligible participants and assessors were unaware of the assignment order. Both the physician and participants will be unaware of the group allocation. Participants were allowed to withdraw from the study at any time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laser acupuncture group (Experimental): This study will use the Handylaser Trion laser manufactured by RJ Laser, Germany.
  It will be used for 40 seconds to deliver 6 J of energy as a pulsed wave (Noiger E) at each acupoint near palms or plantar, such as bilateral LI 4, PC6, KI 3, LR 3.
  For distal points in the four limbs, the laser will be used for 40 seconds at each acupoint to deliver 6J of energy as a pulsed wave (Noiger B), such as bilateral LI11, GB 34, ST 36, SP 6.
  Interventions: Device: laser acupuncture
- sham laser acupuncture group (Sham Comparator): This study will use the sham Handylaser Trion laser manufactured by RJ Laser, without any laser beam delivering. The acupoints of the sham-laser acupuncture are the same as those of the laser acupuncture group.
  Interventions: Device: sham laser acupuncture

INTERVENTIONS:
Device: laser acupuncture — This study will use the Handylaser Trion laser manufactured by RJ Laser, Germany.
  Arms: laser acupuncture group
Device: sham laser acupuncture — This study will use the sham Handylaser Trion laser manufactured by RJ Laser, Germany,and without any laser beam delivering
  Arms: sham laser acupuncture group

SUMMARY:
Diabetic peripheral neuropathy (DPN) is one of the microvascular complications of diabetes mellitus. This can lead to painful and costly clinical sequelae such as foot ulcers, amputation, and neuropathic pain. There are several novel diagnostic methods available for complementary to clinical assessment and may help in the early detection of DPN. However, treatments for DPN and painful DPN are limited.

We will conduct a pilot, single-center, randomized controlled trial in patients with DPN to verify the effect of the laser acupuncture on DPN. With designed inclusion and exclusion criteria, 30 eligible participants will be randomized with 1:1 allocation ratio to the following two groups:(1) the laser acupuncture group (N=15), (2) the sham laser acupuncture group (N=15). Each participant will receive 24 interventions within 8 weeks, three times per week. Participants follow the laser acupuncture protocol in our study. All participants will be clinically assessed by (1) Michigan Neuropathy Screening Instrument (MNSI), (2) questionnaires (BPI(SF)-DPN) for diabetic neuropathic pain assessment, and (3) nerve conduction test.

This research project will validate our novel preliminary findings demonstrating neuroprotective effects of laser acupuncture treatment. Importantly, our data are expected to elucidate how laser acupuncture induces neuroprotection in the clinical setting and provide a scientific base for developing new approaches in the treatment of DPN.

DETAILED DESCRIPTION:
This prospective, randomized, single-center, parallel-group study will be cooperatively conducted in the neurology and traditional Chinese medicine department of Tainan Municipal An-Nan Hospital, China Medical University in Tainan, Taiwan. Study approval will be applied from the TMANH Research Ethics Committee. After screening eligibility and completing baseline assessments, we obtained informed consent from all patients before enrollment. Participants were randomized to either the laser acupuncture, the sham laser acupuncture group using a block randomization method with allocation ratio of 1:1(Figure 7). Before study commencement, the statistician created a randomization sequence using IBM® SPSS® Statistics and contained it in sealed envelopes. The balanced sample size was ensured by dividing the participants into blocks of two. All eligible participants and assessors were unaware of the assignment order. Both the physician and participants will be unaware of the group allocation. Participants were allowed to withdraw from the study at any time.

• Patient eligibility

We included the patients with the following inclusion criteria(Dietzel, et al. 2021):

1. female or male patients (aged over 18 years) with diabetes mellitus type II.
2. patients have symptoms (numbness, tingling, burning, stabbing, shooting pain, etc.) and signs (symmetric decreased distal sensation, or decreased or absent ankle reflexes) of diabetic neuropathy.
3. presence of abnormal nerve conduction study, or presence of neuropathy is likely tested by Semmes-Weinstein 10-g monofilament, or decreased vibration sensation tested by 128Hz vibration tuning fork
4. patients who have completed titration of pain medication or stopped accepting physical therapy against DPN;
5. must provide written informed consent.

The main exclusion criteria for the patients are as follows:

1. severe DPN with muscular weakness of the proximal leg muscles;
2. neuropathy due to other reasons (such as HIVD, malignancy, severe renal disease, hepatitis, thyroid disease, vitamine B12 deficiency, virus infection (such as: human immunodeficiency virus infection, etc), syphilis, alcohol, neurotoxic drug use, inflammatory disease (such as chronic inflammatory demyelinating polyneuropathy), heavy metal intoxication, hereditary disease, etc)
3. severe peripheral artery disease in Fontaine stage IV(Focal tissue necrosis, ulceration or gangrene);
4. traumatic lesions of the nerves or vessels in the lower extremities;
5. opioid use before inclusion in the study;
6. regular use of cannabis or cannabinoids;
7. severe mental illness;
8. severe impairment of cognitive function;
9. pregnancy or lactation
10. obesity (BMI>35 kg/m2); • Randomization and Intervention After screening for inclusion/exclusion criteria, eligible participants signed the written informed consent and completed the baseline assessments that included a quantitative sensory test using the SWM and patient-reported outcome measurements, and the nerve conduction study. Eligible participants completed the baseline assessments within seven days before the interventions.

According to the previous randomization assignment, each patient will be assigned to 2 groups: (1) the laser acupuncture group and (2) the sham laser acupuncture group. Only the statistician aware of the randomized order for each participant. Each participant will receive 24 interventions within 8 weeks, including three interventions per week for 8 weeks. The selected acupoints for laser acupuncture and electro-acupuncture were the same real acupoints, including bilateral LI 4, PC6, LI11, GB 34, ST 36, SP 6, KI 3, LR 3。

• Statistical analysis All data will be analyzed using IBM® SPSS® Statistics version 22 (Statistical Product and Service Solutions Statistics, I.B.M., Inc., Armonk, NY, USA). For demographic data, continuous data will be analyzed using a two-sample t-test or Mann-Whitney U test, while categorical data will be analyzed using Fisher's exact test. If the data of each group fail to pass the Shapiro-Wilk normal distribution test (all p value < 0.05), the between-group differences will be examined using the nonparametric Mann-Whitney U test, and the intra-group differences will be examined using the Wilcoxon signed-rank test. If the measurements of the baseline values will be as per the Shapiro-Wilk normal distribution test (all p value > 0.05), the difference between groups will be examined using a two-sample t-test, and the intra-group difference was examined using a paired t-test. Differences between or within groups were considered significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. female or male patients (aged over 18 years) with diabetes mellitus type II.
2. patients have symptoms (numbness, tingling, burning, stabbing, shooting pain, etc.) and signs (symmetric decreased distal sensation, or decreased or absent ankle reflexes) of diabetic neuropathy.
3. presence of abnormal nerve conduction study, or presence of neuropathy is likely tested by Semmes-Weinstein 10-g monofilament, or decreased vibration sensation tested by 128Hz vibration tuning fork
4. patients who have completed titration of pain medication or stopped accepting physical therapy against DPN;
5. must provide written informed consent.

Exclusion Criteria:

1. severe DPN with muscular weakness of the proximal leg muscles;
2. neuropathy due to other reasons (such as HIVD, malignancy, severe renal disease, hepatitis, thyroid disease, vitamine B12 deficiency, virus infection (such as: human immunodeficiency virus infection, etc), syphilis, alcohol, neurotoxic drug use, inflammatory disease (such as chronic inflammatory demyelinating polyneuropathy), heavy metal intoxication, hereditary disease, etc)
3. severe peripheral artery disease in Fontaine stage IV(Focal tissue necrosis, ulceration or gangrene);
4. traumatic lesions of the nerves or vessels in the lower extremities;
5. opioid use before inclusion in the study;
6. regular use of cannabis or cannabinoids;
7. severe mental illness;
8. severe impairment of cognitive function;
9. pregnancy or lactation
10. obesity (BMI>35 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
the Brief Pain Inventory-Short Form | BPI-SF will be assessed at the baseline
  The primary endpoint was the mean of mean change in the average pain severity between groups. The two arms will measure the average pain severity score of the Brief Pain Inventory-Short Form(Ger, et al. 1999) (BPI-SF) at the 4th week. The BPI-SF average pain severity score uses a 0-10 scale for subject ratings. The items range from 0 to 10 (0 = no pain; 10 = worst pain). The higher the pain severity scores, the worse the degree of pain experienced by the patient. The BPI-SF also measures the pain interference on seven daily functions during the past 24 h, including general activities, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Using numeric scales, the items range from 0 to 10 (0 = no interference; 10= interferes completely). This study will measure the average pain severity and seven pain interference domains for eligible participants.
the Brief Pain Inventory-Short Form | BPI-SF will be assessed at the 4th week
  The primary endpoint was the mean of mean change in the average pain severity between groups. The two arms will measure the average pain severity score of the Brief Pain Inventory-Short Form(Ger, et al. 1999) (BPI-SF) at the 4th week. The BPI-SF average pain severity score uses a 0-10 scale for subject ratings. The items range from 0 to 10 (0 = no pain; 10 = worst pain). The higher the pain severity scores, the worse the degree of pain experienced by the patient. The BPI-SF also measures the pain interference on seven daily functions during the past 24 h, including general activities, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Using numeric scales, the items range from 0 to 10 (0 = no interference; 10= interferes completely). This study will measure the average pain severity and seven pain interference domains for eligible participants.
the Brief Pain Inventory-Short Form | BPI-SF will be assessed at the 8th week
  The primary endpoint was the mean of mean change in the average pain severity between groups. The two arms will measure the average pain severity score of the Brief Pain Inventory-Short Form(Ger, et al. 1999) (BPI-SF) at the 4th week. The BPI-SF average pain severity score uses a 0-10 scale for subject ratings. The items range from 0 to 10 (0 = no pain; 10 = worst pain). The higher the pain severity scores, the worse the degree of pain experienced by the patient. The BPI-SF also measures the pain interference on seven daily functions during the past 24 h, including general activities, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Using numeric scales, the items range from 0 to 10 (0 = no interference; 10= interferes completely). This study will measure the average pain severity and seven pain interference domains for eligible participants.

SECONDARY OUTCOMES:
The Michigan Neuropathy Screening Instrument (MNSI) | MNSI will be assessed at the baseline
  The Michigan Neuropathy Screening Instrument (MNSI) is designed to screen for the presence of diabetic neuropathy. The first part of the screening instrument, the history questionnaire, consists of 15 self-administered "yes or no" questions on foot sensation including pain, numbness and temperature sensitivity. A higher score (out of a maximum of 13 points) indicates more neuropathic symptoms. The second part of the MNSI is a brief physical assessment (completed by health professionals) involving:1) inspection of the feet for deformities, dry skin, hair or nail abnormalities, callous or infection; 2) semi-quantitative assessment of vibration sensation at the dorsum of the great toe; 3) grading of ankle reflexes and 4) monofilament testing. Patients screening positive on the clinical portion of the MNSI (greater than 2 points on a 10 point scale) are considered neuropathic and referred for further evaluation.
The Michigan Neuropathy Screening Instrument (MNSI) | MNSI will be assessed at the 8th week
  The Michigan Neuropathy Screening Instrument (MNSI) is designed to screen for the presence of diabetic neuropathy. The first part of the screening instrument, the history questionnaire, consists of 15 self-administered "yes or no" questions on foot sensation including pain, numbness and temperature sensitivity. A higher score (out of a maximum of 13 points) indicates more neuropathic symptoms. The second part of the MNSI is a brief physical assessment (completed by health professionals) involving:1) inspection of the feet for deformities, dry skin, hair or nail abnormalities, callous or infection; 2) semi-quantitative assessment of vibration sensation at the dorsum of the great toe; 3) grading of ankle reflexes and 4) monofilament testing. Patients screening positive on the clinical portion of the MNSI (greater than 2 points on a 10 point scale) are considered neuropathic and referred for further evaluation
Semmes-Weinstein Monofilament(SWM) | SWM will be assessed at the baseline
  SWM is a clinically easy-to-administer, quantifiable, and reliable tool for evaluating protective sensation loss(Kamei, et al. 2005). Measurements were performed using a set of 20 von Frey monofilaments (Semmes-Weinstein von Frey Aesthesiometer, Stoelting Co., Wood Dale, IL, USA), with evaluator size/target forces ranging from 1.65/0.008 g to 6.65/300 g. Each monofilament was calibrated to a target force in grams (g) within a 5% standard deviation. Measurement sites included the sole, tip of the big toe, palm, and tip of the middle finger. All tests were performed by an independent assessor who was blinded to the allocation of randomization. All the procedures followed the operation manual provided by the filament manufacturer.
Semmes-Weinstein Monofilament(SWM) | SWM will be assessed at the 8th week
  SWM is a clinically easy-to-administer, quantifiable, and reliable tool for evaluating protective sensation loss(Kamei, et al. 2005). Measurements were performed using a set of 20 von Frey monofilaments (Semmes-Weinstein von Frey Aesthesiometer, Stoelting Co., Wood Dale, IL, USA), with evaluator size/target forces ranging from 1.65/0.008 g to 6.65/300 g. Each monofilament was calibrated to a target force in grams (g) within a 5% standard deviation. Measurement sites included the sole, tip of the big toe, palm, and tip of the middle finger. All tests were performed by an independent assessor who was blinded to the allocation of randomization. All the procedures followed the operation manual provided by the filament manufacturer.
Nerve conduction velocity (NCV) | NCV will be assessed at the baseline
  NCV will be performed on both lower extremities at baseline and the week 8 (the end of treatment). Peroneal motor nerve conduction velocity (MNCV), sural sensory nerve conduction velocity (SNCV), and tibial motor nerve conduction velocity (MNCV) will be measured.
Nerve conduction velocity (NCV) | NCV will be assessed at the 8th week
  NCV will be performed on both lower extremities at baseline and the week 8 (the end of treatment). Peroneal motor nerve conduction velocity (MNCV), sural sensory nerve conduction velocity (SNCV), and tibial motor nerve conduction velocity (MNCV) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hung Chen, PhD, Principal Investigator — China Medical University, China
Locations (1):
- Tainan Municipal An Nan Hospital-China Medical University, Tainan, Taiwan